CLINICAL TRIAL: NCT02186834
Title: Investigator-Initiated Phase I/II Clinical Trial of Selinexor (KPT-330) and Liposomal Doxorubicin for Relapsed and Refractory Multiple Myeloma
Brief Title: Selinexor (KPT-330) and Liposomal Doxorubicin For Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17814
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Refractory; Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Neoplasms, Plasma Cell | interventions — selinexor; liposomal doxorubicin; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selinexor, Liposomal Doxorubicin and Dexamethasone (Experimental): Combination Therapy: Phase I Dose Escalation followed by Phase 2 treatment at Recommended Phase 2 Dose (RP2D).
  After the initial screening visit and registration in the study, participants will receive Selinexor orally at a dose of 80 mg along with dexamethasone for 1 day. One week later, patients will receive weekly selinexor at a starting dose from 60 mg once a week to 80 mg twice a week in combination with pegylated liposomal doxorubicin at a starting dose of 20 mg/m², and dexamethasone 40 mg orally weekly.
  Interventions: Drug: Selinexor; Drug: Liposomal doxorubicin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Selinexor orally as outlined in the study treatment arm.
  Other Names: KPT-330
Drug: Liposomal doxorubicin — Pegylated liposomal doxorubicin at a starting dose of 20 mb/m² as outlined in the treatment arm.
  Other Names: Lipodox; LD
Drug: Dexamethasone — Participants will be instructed to take Dexamethasone 40 mg (10 tablets) orally once weekly with meals (ideally with breakfast to minimize insomnia). Participants older than 75 years and patients previously intolerant to 40 mg dosage will be allowed to receive 20 mg (5 tablets) once a week.
  Other Names: Decadron

SUMMARY:
The main purpose of this study is to determine the recommended doses of selinexor in combination with liposomal doxorubicin and dexamethasone for patients with relapsed and refractory myeloma. In addition, the study will assess whether this combination with effective for patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed and refractory multiple myeloma who have received at least 2 prior therapies which must include lenalidomide and a proteasome inhibitor. Patients must have disease refractory to the most recent therapy. Refractory myeloma is defined as progressive disease during or within 60 days of last therapy. Patients must have previously received or be ineligible for (or refused) autologous stem cell transplant.
* Must have measurable myeloma paraprotein levels in serum (≥ 0.5 g/dL) or urine (≥ 0.2 g excreted in a 24-hour urine collection sample) or by free light chain (involved free light chain greater than 100 mg/L).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. ECOG 2 allowed if due to bone disease
* Must have an echocardiogram or multigated acquisition (MUGA) scan indicating left ventricular ejection fraction (LVEF) ≥ 50% within 42 days prior to first dose of study drug
* Adequate hematological function
* Adequate hepatic function within 14 days prior to loading phase (day -14)
* Adequate renal function within 14 days prior to loading: estimated creatinine clearance of ≥ 30 mL/min, (Cockcroft and Gault)
* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening. Male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.

Exclusion Criteria:

* Women who are pregnant or lactating
* Radiation, chemotherapy, or immunotherapy or any other approved anticancer therapy ≤2 weeks prior to day -7 (beginning of loading phase)
* Major surgery within four weeks before Day -7
* Myocardial infarct within 6 months before enrollment, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
* Prior cumulative exposure to doxorubicin (including liposomal preparation) > 350mg/m^2
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; patients with controlled infection or on prophylactic antibiotics are permitted in the study
* Known to be HIV seropositive
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) RNA or HBsAg (HBV surface antigen)
* Any underlying condition that would significantly interfere with the absorption of an oral medication
* Grade >2 peripheral neuropathy at baseline (within 14 days prior to loading phase (day -7))
* Serious psychiatric or medical conditions that could interfere with treatment
* Participation in an investigational anti-cancer study within 3 weeks prior to day -7(beginning of loading phase)
* Concurrent therapy with approved or investigational anticancer therapeutic
* Coagulation problems and active bleeding in the last month
* Previous allogeneic transplant within 6 months and have evidence of clinically significant graft versus host disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2018-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachid Baz, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan

REFERENCES:
- [Derived] Turner JG, Dawson JL, Grant S, Shain KH, Dalton WS, Dai Y, Meads M, Baz R, Kauffman M, Shacham S, Sullivan DM. Treatment of acquired drug resistance in multiple myeloma by combination therapy with XPO1 and topoisomerase II inhibitors. J Hematol Oncol. 2016 Aug 24;9(1):73. doi: 10.1186/s13045-016-0304-z. PMID 27557643

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center and Karmanos Cancer Center September 2014 through May 2017.
Pre-assignment Details: 6 of the 14 participants treated at RP2D moved on from Dose 2m arm in the dose escalation portion of study.
Groups:
- Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1: Dose 1: Participants were administered Lipodox 20 mg/m^2 via IV on Day 1 of cycle. Selinexor at 40 mg was given orally on days 1,8 and 15 of the cycle. Dexamethasone at 40 mg was given orally on days 1, 8 and 15.
- Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2: Dose 2: Participants were administered Lipodox 20 mg/m^2 on Day 1 of cycle. Selinexor at 80 mg was given orally on days 1,8 and 15 of the cycle. Dexamethasone at 40 mg was given orally on days 1, 8 and 15.
- Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1m: Dose 1m: Participants were administered Lipodox 20 mg/m^2 on Day 1 of cycle. Selinexor at 60 mg was given orally on days 1,8 and 15 of the cycle. Dexamethasone at 40 mg was given orally on days 1, 8 and 15.
- Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2m: Dose 2m: Participants were administered Lipodox 20mg/m^2 on Day 1 of cycle. Selinexor at 80 mg was given orally on days 1,8 and 15 of the cycle. Dexamethasone at 40 mg was given orally on days 1, 8 and 15.
- Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 3m: Dose 3m: Participants were administered Lipodox 20mg/m^2 on Day 1 of cycle. Selinexor at 80 mg was given orally on days 1,3, 8 and 10 of the cycle. Dexamethasone at 40 mg was given orally on days 1, 8 and 15.
- Selinexor, Liposomal Doxorubicin and Dexamethasone- RP2D: Phase 2 Dose: Participants were administered Lipodox 20 mg/m^2 on Day 1 of cycle. Selinexor at 80 mg was given orally on days 1,8 and 15 of the cycle. Dexamethasone at 40 mg was given orally on days 1, 8 and 15.
Period: Dose Escalation
Arm/Group | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1 | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2 | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1m | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2m | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 3m | Selinexor, Liposomal Doxorubicin and Dexamethasone- RP2D
Started | 6 | 3 | 0 | 7 | 4 | 0
Completed | 6 | 3 | 0 | 6 | 4 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Period: Treatment at RP2D
Arm/Group | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1 | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2 | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1m | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2m | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 3m | Selinexor, Liposomal Doxorubicin and Dexamethasone- RP2D
Started | 0 | 0 | 0 | 0 | 0 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Died prior to treatment | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received treatment
Groups:
- Selinexor, Liposomal Doxorubicin and Dexamethasone: Combination Therapy: Phase I Dose Escalation followed by Phase 2 treatment at Recommended Phase 2 Dose (RP2D)
Arm/Group | Selinexor, Liposomal Doxorubicin and Dexamethasone
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 60 [49 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 21
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D): Selinexor on Days 1, 8 and 15 when given in combination with Lipodox 20 mg/m^2 and Dexamethasone 40 mg.
  Dose level 1: 40 mg in combination with Lipodox and Dexamethasone.
  Dose level 2: 80 mg (D1,8,15) in combination with Lipodox and Dexamethasone.
  Dose level 2m: 80 mg (D1,8,15) in combination with Lipodox and Dexamethasone.
  Dose level 3m: 80 mg (D1,3,8,10) in combination with Lipodox and Dexamethasone.
Time Frame: Up to 12 months
Population: All participants treated during dose escalation
Measure: Number; unit: mg
Arm/Group | Selinexor, Liposomal Doxorubicin and Dexamethasone
Number analyzed (Participants) | 19
mg | 80

2. Primary Outcome: Overall Response Rate (ORR) - All Participants
Description: ORR per the modified uniform response criteria of the International Myeloma Working Group (IMWG), partial response and better. Partial Remission (PR): >/= 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >/= 90% or to < 200 mg per 24 hours; Very Good Partial Remission (VGPR): Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours; Complete Remission (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and </= 5% plasma cells in bone marrow. Stable Disease: Not meeting criteria for CR, VGPR, PR, or progressive disease. Minimal response: Less than 50% decrease in M protein. Not evaluable: Cannot be measured because enough information has not been collected.
Time Frame: Up to 24 months
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor, Liposomal Doxorubicin and Dexamethasone
Number analyzed (Participants) | 27
Participants
  >/= Very Good Partial Response | 2
  >/= Partial Response | 4
  >/= Minimal Response | 9
  Stable Disease | 8
  Not Evaluable | 4

3. Primary Outcome: Overall Response Rate (ORR) -All Participants Treated at Recommended Phase 2 Dose
Description: Determine the overall response rate per the modified uniform response criteria of the International Myeloma Working Group (IMWG), partial response and better. Partial Remission (PR): >/= 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by >/= 90% or to < 200 mg per 24 hours; Very Good Partial Remission (VGPR): Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours; Complete Remission (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and </= 5% plasma cells in bone marrow.
Time Frame: Up to 24 months
Population: All participants treated at recommended phase 2 dose, regardless of when they joined the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor, Liposomal Doxorubicin and Dexamethasone
Number analyzed (Participants) | 14
Participants
  >/= Very Good Partial Response | 0
  >/= Partial Response | 1
  >/= Minimal Response | 2
  Stable Disease | 4
  Not Evaluable | 1

ADVERSE EVENTS:
Time Frame: 3 years, 2 months
Description: All Adverse Events (AEs) and Serious Adverse Events (SAEs) at all grade levels, regardless of causality have been reported in this section. One participant died prior to treatment but after consent. Only participants who received treatment were considered at Risk for Serious and Other Adverse Events.
Arm/Group | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1 | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2 | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1m | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2m | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 3m | Selinexor, Liposomal Doxorubicin and Dexamethasone- RP2D
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/3 | 0/0 | 1/7 | 0/4 | 1/8
Serious Adverse Events (participants affected / at risk) | 4/6 | 1/1 | 0/0 | 6/7 | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 5/6 | 3/3 | 0/0 | 7/7 | 4/4 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1 (N=6) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2 (N=1) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1m (N=0) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2m (N=7) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 3m (N=4) | Selinexor, Liposomal Doxorubicin and Dexamethasone- RP2D (N=7)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystitis pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RSV pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1 (N=6) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2 (N=3) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 1m (N=0) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 2m (N=7) | Selinexor, Liposomal Doxorubicin and Dexamethasone- Dose 3m (N=4) | Selinexor, Liposomal Doxorubicin and Dexamethasone- RP2D (N=7)
Nausea (Gastrointestinal disorders) | 4 (6) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (6) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (6) | 1 (2) | 0 (0) | 2 (4) | 1 (1) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (10) | 3 (12) | 0 (0) | 3 (5) | 1 (1) | 1 (3)
White blood cell decreased (Investigations) | 5 (10) | 3 (9) | 0 (0) | 3 (4) | 1 (3) | 0 (0)
Neurtrophil count decreased (Investigations) | 4 (9) | 3 (5) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CPK increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (4) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Fever (General disorders) | 1 (3) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders - Other (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5) | 2 (3) | 0 (0) | 2 (5) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (7) | 3 (8) | 0 (0) | 3 (3) | 2 (3) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic thrombocytopenia purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorders -Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders -Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmer-plantar erythrodesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT02186834/Prot_SAP_000.pdf